CLINICAL TRIAL: NCT04817618
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Iptacopan (LNP023) in Complement 3 Glomerulopathy.
Brief Title: Study of Efficacy and Safety of Iptacopan in Patients With C3 Glomerulopathy.
Acronym: APPEAR-C3G
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLNP023B12301; 2020-004589-21 (EudraCT Number)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: C3G
Keywords: LNP023; iptacopan; C3G; UPCR; eGFR; proteinuria; Quality of life
MeSH Terms: conditions — Proteinuria | interventions — iptacopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iptacopan 200mg (Experimental): iptacopan 200 mg b.i.d.
  Interventions: Drug: iptacopan
- Placebo to iptacopan 200mg (Placebo Comparator): Placebo to iptacopan 200mg b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to iptacopan 200mg b.i.d. (Adults 200mg b.i.d; Adolescents 2x 100mg b.i.d)
  Arms: Placebo to iptacopan 200mg
Drug: iptacopan — iptacopan 200 mg b.i.d. (Adults 200mg b.i.d; Adolescents 2x 100mg b.i.d)
  Other Names: LNP023
  Arms: iptacopan 200mg

SUMMARY:
The Primary Completion Date and Study Completion Date have been updated to reflect completion of the adolescent cohort, which has been added to the protocol.

The study is designed as a multicenter, randomized, double-blind, parallel group, placebo-controlled study to evaluate the efficacy and safety of iptacopan (LNP023) in complement 3 glomerulopathy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of iptacopan compared to placebo and standard of care in patients with native C3G. CLNP023B12301 is a Phase 3 pivotal trial for registration of iptacopan in C3G. The study aims to determine the reduction in UPCR and improvement in eGFR in participants treated with iptacopan compared to placebo, as well as the proportion of participants who achieve a composite renal endpoint consisting of eGFR and UPCR elements. These effects of iptacopan in conjunction with increases in serum C3 levels will provide support for an iptacopan profile that includes stabilization of eGFR, clinically meaningful reductions in proteinuria and inhibition of the complement AP. Kidney biopsies will be performed in adult participants to evaluate histopathological improvements in immunofluorescence and light microscopy that support these functional benefits of iptacopan.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants age ≥ 12 and ≤ 60 years at screening.
* Diagnosis of C3G as confirmed by renal biopsy within 12 months prior to enrollment in adults and within 3 years in adolescents.
* Prior to randomization, all participants must have been on a maximally recommended or tolerated dose of an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) for at least 90 days. The doses of other antiproteinuric medications including mycophenolic acid, corticosteroids and mineralocorticoid receptor antagonists should be stable for at least 90 days prior to randomization.
* Reduced serum C3 (defined as less than 0.85 x lower limit of the central laboratory normal range) at Screening.
* UPCR ≥ 1.0 g/g sampled from the first morning void urine sample at Day -75 and Day -15.
* Estimated GFR (using the CKD-EPI formula for ages ≥ 18 years and modified Schwartz formula for ages 12 to 17 years) or measured GFR ≥ 30 ml/min/1.73m2 at screening and Day -15.
* Mandatory vaccination against Neisseria meningitidis and Streptococcus pneumoniae prior to the start of study treatment.
* If not previously vaccinated or if a booster is required, vaccination against Haemophilus influenzae infections should be given, if available and according to local regulations, at least 2 weeks prior to the first study treatment administration. If study treatment has to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment should be initiated.

Exclusion Criteria:

* Participants who have received any cell or organ transplantation, including a kidney transplantation.
* Rapidly progressive crescentic glomerulonephritis defined as a 50% decline in the eGFR within 3 months with renal biopsy findings of glomerular crescent formation seen in at least 50% of glomeruli.
* Renal biopsy showing interstitial fibrosis/tubular atrophy (IF/TA) of more than 50%
* Monoclonal gammopathy of undetermined significance (MGUS) confirmed by the measurement of serum free light chains or other investigation as per local standard of care.
* Participants with an active systemic bacterial, viral or fungal infection within 14 days prior to study treatment administration
* The presence of fever ≥ 38°C (100.4°F) within 7 days prior to study treatment administration.
* A history of recurrent invasive infections caused by encapsulated organisms, e.g., N. meningitidis and S. pneumoniae.
* The use of inhibitors of complement factors (e.g., Factor B, Factor D, C3 inhibitors, anti C5 antibodies, C5a receptor antagonists) within 6 months prior to the Screening visit.
* The use of immunosuppressants (except mycophenolic acids), cyclophosphamide or systemic corticosteroids at a dose >7.5 mg/day (or equivalent for a similar medication) within 90 days of study drug administration.
* Acute post-infectious glomerulonephritis at screening based upon the opinion of the investigator.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Adult cohort: Log-transformed ratio to baseline in UPCR (sampled from a 24-hour urine collection) | 6 months (double-blind)
  To demonstrate the superiority of iptacopan compared to placebo in reducing proteinuria at 6 months of treatment.
Adolescent cohort: Log-transformed ratio to baseline in UPCR (sampled from a 24-hour urine collection) | 6 months (double-blind)
  To evaluate the effect of iptacopan on proteinuria at 6 months.
Change from baseline in log-transformed UPCR at the 12-month visit (both study treatment arms). | 12 months (double-blind and open-label)
  To evaluate the effect of iptacopan on proteinuria at 12 months.
Change in log-transformed UPCR from the 6-month visit to the 12-month visit in the placebo arm | From month 6 to month 12 (open-label)
  To evaluate the effect of iptacopan on proteinuria at 12 months.

SECONDARY OUTCOMES:
Change from baseline in eGFR. | 6 months (double-blind)
  To demonstrate the superiority of iptacopan vs. placebo in improving eGFR.
Proportion of participants who meet the criteria for achieving a composite renal endpoint | 6 months (double-blind)
  To demonstrate the superiority of iptacopan vs. placebo in the proportion of participants who meet the criteria for achieving a composite renal endpoint.
  A participant meets the requirements of the composite renal endpoint if he/she satisfies: (1) a stable or improved eGFR compared to the baseline visit (≤15% reduction in eGFR), and (2) a ≥50% reduction in UPCR compared to the baseline visit.
Adult cohort: Change from baseline in disease total activity score in a renal biopsy. | 6 months (double-blind)
  To demonstrate the effect of iptacopan vs placebo in reducing glomerular inflammation in the kidney.
Change from baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score. | 6 months (double-blind)
  To assess the effect of iptacopan compared to placebo in improvement of patient reported fatigue.
Number of participants with abnormal clinically significant vital signs, ECGs and safety laboratory measurements | 6 months (double-blind)
  To evaluate the safety and tolerability of iptacopan compared to placebo.
Number of participants with study drug discontinuation due to an AE | 6 months (double-blind)
  To evaluate the safety and tolerability of iptacopan compared to placebo
Proportion of participants who meet the criteria for achieving a composite renal endpoint | 12 months (double-blind and open-label)
  To evaluate the effect at 12 months of iptacopan on a composite renal endpoint. A participant meets the requirements of the composite renal endpoint if he/she satisfies: (1) a stable or improved eGFR compared to the baseline visit (≤15% reduction in eGFR), and (2) a ≥50% reduction in UPCR compared to the baseline visit.
Proportion of patients achieving a composite renal endpoint from the 6-month visit to the 12-month visit of the placebo arm | month 6, month 12 (open-label)
  To evaluate the effect at 12 months of iptacopan on a composite renal endpoint. A participant meets the requirements of the composite renal endpoint if he/she satisfies: (1) a stable or improved eGFR compared to the baseline visit (≤15% reduction in eGFR), and (2) a ≥50% reduction in UPCR compared to the 6 months visit.
Change from baseline in the total activity score in a renal biopsy at 12 months | Baseline, month 12 (double-blind and open-label)
  To evaluate the effect at 12 months of iptacopan in reducing glomerular inflammation in the kidney.
Change in the total activity score in a renal biopsy from the 6-month visit to the 12-month visit of the placebo arm. | month 6, month 12 (open-label)
  To evaluate the effect at 12 months of iptacopan in reducing glomerular inflammation in the kidney.
Change from baseline in the FACIT-Fatigue score at 12 months | Baseline, month 12 (double-blind and open-label)
  To evaluate the effect at 12 months of iptacopan in improvement of patient reported fatigue
Change in the FACIT-Fatigue score from the 6-month visit to the 12-month visit of the placebo arm | month 6, month 12 (open-label)
  To evaluate the effect at 12 months of iptacopan in improvement of patient reported fatigue
Number of participants with abnormal clinically significant vital signs, ECGs and safety laboratory measurements | 12 months (double-blind and open-label)
  To evaluate the safety and tolerability of iptacopan during the 6-month open-label treatment period as well as the entire 12- month treatment period
Number of participants with study drug discontinuation due to an AE | 12 months (double-blind and open-label)
  To evaluate the safety and tolerability of iptacopan during the 6-month open-label treatment period as well as the entire 12- month treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- United States (9):
  - Childrens Hospital Colorado, Aurora, Colorado
  - Nicklaus Childrens Hospital, Miami, Florida
  - Georgia Nephrology Research Inst, Lawrenceville, Georgia
  - University of Iowa Health Care, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - Albany Medical Center, Albany, New York
  - Col Uni Med Center New York Presby, New York, New York
  - Baylor Scott and White Research, Temple, Texas
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Belgium (2):
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
- Brazil (7):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Pernambuco, Recife
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Wuhan
- Novartis Investigative Site, Prague, Czechia
- France (4):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Mainz
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion Crete
  - Novartis Investigative Site, Thessaloniki
- India (5):
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (3):
  - Novartis Investigative Site, Ranica, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Niigata
- Netherlands (2):
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Nijmegen
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Port de Sagunt, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Talas Kayseri
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kavanagh D, Bomback AS, Vivarelli M, Nester CM, Remuzzi G, Zhao MH, Wong EKS, Wang Y, Krishnan I, Schuhmann I, Trapani AJ, Webb NJA, Meier M, Israni RK, Smith RJH; APPEAR-C3G investigators. Oral iptacopan therapy in patients with C3 glomerulopathy: a randomised, double-blind, parallel group, multicentre, placebo-controlled, phase 3 study. Lancet. 2025 Oct 11;406(10512):1587-1598. doi: 10.1016/S0140-6736(25)01148-1. Epub 2025 Sep 25. PMID 41016405